CLINICAL TRIAL: NCT03850470
Title: The Diagnostic Accuracy of the Clinical Examination in Common Musculoskeletal Pathologies
Brief Title: The Diagnostic Accuracy of the Clinical Examination
Status: Terminated | Type: Observational
Why Stopped: PI left the institution
Sponsor: High Point University (Other)
Responsible Party: Sponsor
Other Study IDs: 201802-695
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Musculoskeletal Pain; Musculoskeletal Injury
Keywords: Diagnostic accuracy; Clinical examination; neck; back; shoulder; hip; knee; foot; ankle; stress fracture
MeSH Terms: conditions — Musculoskeletal Pain; Fractures, Stress | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Musculoskeletal Pain: Subjects reporting for care with complaints of musculoskeletal pain will be examined and a diagnosis and plan of care will be established. The accuracy of the clinical examination will be compared to pathology detected by MRI
  Interventions: Diagnostic Test: clinical examination; Other: MRI

INTERVENTIONS:
Diagnostic Test: clinical examination — Thorough examination including history, screening, motion testing, strength testing, special testing
Other: MRI — Low field MRI .25 Tesla

SUMMARY:
This study examines the diagnostic accuracy of the clinical examination as compared to MRI findings

DETAILED DESCRIPTION:
When patients get musculoskeletal pain and seek care, the healthcare professional performs a detailed clinical examination to determine a diagnosis and determine a plan of care which often includes imaging. There are only a few studies that have looked at the accuracy of the clinical examination in a primary care setting, most studies having been performed in a specialty practice treating Orthopedic or Sports injuries. In these practices, surgery has become and remains the gold standard. However, in primary care, often imaging like Magnetic Resonance Imaging (MRI) has become the the criterion standard. This double blind study will compare the diagnosis reached by clinical exam to the results found on MRI. In addition, the examining clinician will report their recommended plan of care after the examination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18-80 years old with musculoskeletal pain/dysfunction

Exclusion Criteria:

* Outside the inclusion age range, pain/dysfunction of other than musculoskeletal origin, those in whom MRI is contraindicated for example, with shrapnel in the body

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These will be patients with musculoskeletal pain or dysfunction that report to one of our several clinics as a normal part of procedure
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
likelihood ratios | 5 years
  combination of sensitivity
Area under the curve | 5 years
  measure of accuracy of the clinical exam

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Hegedus, PhD, Principal Investigator — Professor
Locations (1):
- High Point University, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared only with those submitted to and approved by our IRB. There are no plans to share any data outside of our research group